CLINICAL TRIAL: NCT05034445
Title: A Prospective Study of Advanced NSCLC Patients Genomic Landscape Through Sputum NGS Detection
Brief Title: Whether Sputum Can Serve as an Alternative Source for Liquid Biopsy in Patients With Lung Cancer
Status: Completed | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Director, Guangzhou Institute of Respiratory Disease
Other Study IDs: CROC2004
Record Dates: First submitted 2021-07-12; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tumor DNA obtained from patients' tissue biopsy, plasma or sputum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sputum group: Sputum samples from more than 30 newly diagnosed advanced NSCLC patients with 520 Panel sequencing (sputum 1000X)
  Interventions: Diagnostic Test: Next generation sequencing
- Tissue group: Clinical data review to obtain corresponding tissue samples from more than 30 newly diagnosed advanced NSCLC patients with 520 Panel sequencing (tissue 1000X)
- Plasma group: Clinical data review to obtain corresponding plasma samples from more than 30 newly diagnosed advanced NSCLC patients with 520 Panel sequencing (plasma 10000X)

INTERVENTIONS:
Diagnostic Test: Next generation sequencing — Extract DNA from sputum sample, minimum DNA amount should be over 50ng.
  Groups: Sputum group

SUMMARY:
This study intends to use Onconscreen plus 520 Panel (Burning Rock, China) to conduct NGS testing in sputum, tissues and blood samples of patients with advanced NSCLC. In order to explore the use of sputum as a diagnosis method for NSCLC patients, we will collect relevant clinical information and follow-up treatment information. The primary endpoint will reveal the effectiveness, accuracy, and feasibility in sputum, as compared to tissues and blood samples. This study aims to study the feasibility and advantages/disadvantages of using sputum as an noval body fluid biopsy option.

DETAILED DESCRIPTION:
With the advancements in the development of targeted therapy, the detection of actionable genes has become routine practice in diagnosing lung cancer, especially in non-small cell lung cancer (NSCLC). Due to its non-invasiveness and great accessibility, plasma-based mutation profiling, with a sensitivity of approximately 70% relative to tissue samples, is widely used in clinical settings. Profiling using other body fluids such as pleural effusion, ascites, cerebrospinal fluid have been actively explored. Circulating cell-free DNA has also been shown to be present in other bodily fluids such as sputum and urine, which have potential to serve as liquid biopsy media for comprehensive mutation profiling. In this study, we investigated the potential of sputum obtained from NSCLC patients for mutation profiling using matched tissue, plasma and sputum from more than 30 advanced-stage NSCLC patients.

Baseline tissues, plasma and sputum samples from more than 30 newly diagnosed advanced NSCLC patients with 520 Panel sequencing (tissue 1000X, sputum 1000X, plasma cfDNA 10000X), in different methods will be compared.

Primary endpoints:

1、Compare different sample types with concordence rate, sensitivity, and specificity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage IIIB-IV NSCLC in AJCC TNM stage (8th edition) confirmed with histology or cytology;
2. Newly diagnosed;
3. There are sufficient samples that meet the requirements for examination;
4. Eligible for the next anti-tumor systemic treatment;
5. Willing to sign the consent inform, age ≥18 years;
6. Patients willing to cooperate with the planned follow-up schedule;
7. Permit to collect clinical data needed by the institute.

Exclusion Criteria:

1. Diagnosed with other malignant tumors at the same time (except for fully treated cervical carcinoma in situ, basal or squamous cell skin cancer);
2. The patient has other serious diseases that may affect follow-up and short-term survival;
3. Any other medical conditions and social/psychological problems that investigator evaluated is not suitable to enroll in this study;
4. Absents of contrast-enhanced magnetic resonance imaging (MRI) or contrast-enhanced computer tomography (CT) during clinical follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planning to enroll more than 30 newly diagnosed advanced NSCLC patients, age over 18 years old following the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Compare different sample types with concordence rate, sensitivity, and specificity. | up to 2 years
  1. Concordance rate was defined as the fraction of the total number of true positive and true negative patients relative to the cohort or indicated subgroup;
  2. Sensitivity rate means true positive rate, true positive patients were defined as those who carried at least one genomic alteration that were detected in both matched samples.
  3. Specificity rate means ture negative rate, patients were as defined true negative if no alteration was detected from either matched sample.

CONTACTS AND LOCATIONS:
Overall Officials: Chengzhi Zhou, Dr. PhD., Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Zhou Chengzhi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided